CLINICAL TRIAL: NCT05928598
Title: Drug-Resistant Epilepsy (DRE) Goals for Epilepsy Clinical Visits mHealth Epilepsy Visit Planner Trial
Brief Title: Goals for Epilepsy Clinic Visits Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Chloe Hill, Assistant Professor of Neurology, University of Michigan
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00231921; K23NS126495-02 (NIH)
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Drug Resistant Epilepsy
Keywords: Survey; Quality of life; Communication tool; Patient-provider communication
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Enrollment for the trial will include 76 participants for the standard care arm and will include 76 participants for the intervention arm (who will receive the Epilepsy Visit Planner). The study team will enroll for the standard arm and then for the intervention arm for an approximate total of 152 participants. Additionally, approximately 10 providers will be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard care arm - patient participants (Other): This group will be enrolled first.
  Interventions: Behavioral: Survey questionnaires
- Intervention arm (Epilepsy Visit Planner) - patient participants (Experimental): This group will be enrolled after the standard care arm enrollment is completed.
  Interventions: Behavioral: Survey questionnaires; Behavioral: Epilepsy Visit Planner
- Intervention arm (Epilepsy Visit Planner) - provider participants (Other): Epilepsy providers will be recruited from the University of Michigan (approximately 10 providers).
  Interventions: Behavioral: Questionnaires for Providers

INTERVENTIONS:
Behavioral: Survey questionnaires — Participants will be enrolled before a scheduled clinic appointment. Following the clinic visit, the research staff will ask the patient to complete questionnaires electronically (or by phone if patient prefers) within three days after the baseline clinic visit and then at three months following this visit. Additionally, some data will be obtained from the participant's medical record.
  Arms: Intervention arm (Epilepsy Visit Planner) - patient participants; Standard care arm - patient participants
Behavioral: Epilepsy Visit Planner — Participants will be identified before a scheduled clinic appointment. Prior to the clinic visit (at the site) the participants will meet with a research staff to obtain written informed consent and then present the Epilepsy Visit Planner to the patient. Participants will be encouraged to use the Planner and share the Planner's output with the provider during the clinic visit. In some cases, there could be an option for the participants to consent prior to the visit and have a virtual presentation of the Planner.
  Following the clinic visit, the research staff will ask the participants to complete questionnaires electronically (or by phone if patient prefers) within three days after the baseline clinic visit and then at three months following this visit. Additionally, some data will be obtained from the participant's medical record.
  Arms: Intervention arm (Epilepsy Visit Planner) - patient participants
Behavioral: Questionnaires for Providers — Providers will be asked to complete a survey after the clinic visit for the intervention group.
  Arms: Intervention arm (Epilepsy Visit Planner) - provider participants

SUMMARY:
The purpose of this project is to conduct a trial to assess whether patients that receive a tablet-based waiting room priority communication tool (the "Epilepsy Visit Planner") have improved outcomes compared to patients that do not receive the tool.

The project's hypotheses are:

* Patients that receive the Epilepsy Visit Planner will have improved patient-provider communication compared to the non-planner group.
* Patients that receive the Epilepsy Visit Planner will have improved quality of life scores.
* The Epilepsy Visit Planner will score highly on process measures of feasibility and acceptability, demonstrating suitability for future larger scale study.

Additionally, there is a related survey project that is not part of the clinical trial and will not be included in this registration information.

ELIGIBILITY:
Inclusion Criteria - Patient Participants:

* Adults with drug-resistant epilepsy
* Participants receiving care through the Epilepsy clinics at the University of Michigan

Exclusion Criteria - Patient Participants:

* <18 years old
* Non-English speaking
* Do not clearly have drug-resistant epilepsy
* Moderate-to-severe cognitive impairment that precludes study questionnaire completion

Inclusion Criteria - Provider Participants:

-University of Michigan epilepsy providers

Exclusion Criteria - Provider Participants:

-Not University of Michigan epilepsy providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Efficacy in Patient-Physician Interactions Questionnaire (PEPPI), difference in mean score between trial arms | Baseline
  This is a 10-item measure with Likert scale (range 1-5 for each response) with a score range of 10-50 (higher score indicating higher perceived efficacy in communicating with providers).

SECONDARY OUTCOMES:
Perceived Involvement in Care (PICS), difference in mean score between trial arms | Baseline
  This is a 13-item measure with binary agree/disagree responses (0 points for disagree and 1 point for agree) and higher scores reflecting a greater degree of perceived patient activity and involvement.
Quality of Life in Epilepsy (QOLIE-10) inventory, difference in mean score between trial arms | 3 months after baseline visit
  This is a 10-item measure with Likert scale (range 1-5 for each response) with a score range of 10-50 (lower score indicates better health outcome).
Feasibility, assessed in intervention arm | Baseline - intervention arm only
  Three questions will be asked regarding if the Planner was completed, if the Planner was shared during the visit, and how the Planner impacted visit length. Both patient participants and provider participants will complete these questions.
Acceptability of Intervention Measure, assessed in intervention arm | Baseline - intervention arm only
  There are 4 questions that will be completed by the patient participants and provider participants that evaluate the acceptability of the intervention. The question responses have a Likert scale from 1(completely disagree) to 5 (completely agree). There is a range from 5-25 with a higher score indicating a higher acceptability of the intervention tool.

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Hill, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No